CLINICAL TRIAL: NCT03816839
Title: A Phase 1 Study for the Safety, Efficacy, Pharmacokinetics and Pharmacodynamics Evaluation of SAR439859, Administered Orally as Monotherapy in Japanese Postmenopausal Women With Estrogen Receptor-Positive And Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer (AMEERA-2)
Brief Title: Evaluation of Orally Administered Amcenestrant (SAR439859) in Japanese Postmenopausal Patients With Advanced Breast Cancer (AMEERA-2)
Acronym: AMEERA-2
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to prematurely stop the study, not linked to any safety concern.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TED15954; U1111-1217-2758 (Other: ICTRP)
Record Dates: First submitted 2019-01-17; First posted 2019-01-25 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAR439859 (Experimental): administered orally once daily or twice daily as monotherapy in fasted or fed state
  Interventions: Drug: Amcenestrant (SAR439859)

INTERVENTIONS:
Drug: Amcenestrant (SAR439859) — Pharmaceutical form: Capsules
  Route of administration: Oral

SUMMARY:
Primary Objective:

To assess the incidence rate of dose-limiting toxicity and to confirm the recommended dose as well as the maximum tolerated dose of SAR439859 administered as monotherapy to Japanese postmenopausal women with estrogen receptor positive and human epidermal growth factor receptor 2-negative advanced breast cancer.

Secondary Objective:

* To characterize the overall safety profile of SAR439859 administered as monotherapy.
* To characterize the pharmacokinetic profile of SAR439859 administered as monotherapy.
* To evaluate the antitumor activity of SAR439859 administered as monotherapy and the clinical benefit rate (complete response, partial response and stable disease ≥ 24 weeks).

DETAILED DESCRIPTION:
The duration of the study for an individual participant will include a period to assess eligibility (screening period) of up to 4 weeks (28 days), a treatment period of at least 1 cycle (28 days) of study treatment, and an End of Treatment (EOT) visit at least 30 days (or until the participant receives another anticancer therapy, whichever is earlier) following the last administration of study treatment. Study treatment may continue until precluded by unacceptable toxicity, disease progression, or upon participant's request.

ELIGIBILITY:
Inclusion criteria :

* Participants must be postmenopausal women.
* Breast adenocarcinoma patients with locally advanced not amenable to radiation or surgery, inoperable and/or metastatic disease.
* Either the primary or any metastatic site must be positive for estrogen receptor (ER) (>1% staining by immunohistochemistry).
* Either the primary tumor or any metastatic site must be human epidermal growth factor receptor 2 non-overexpressing.
* Patients with at least 6 months of prior endocrine therapy.

Exclusion criteria:

* Eastern Cooperative Oncology Group Performance Status (ECOG) ≥2.
* Significant concomitant illness that would adversely affect participation in the study.
* Patients with a life expectancy less than 3 months.
* Patient not suitable for participation, whatever the reason.
* Major surgery within 4 weeks prior to first study treatment administration.
* Treatment with strong and moderate cytochrome P450 3A inhibitors/inducers.
* Patients with known endometrial disorders, uterine bleeding or ovarian cysts.
* Treatment with anticancer less than 2 weeks before first study treatment.
* Prior treatment with selective estrogen receptor down (SERD)-regulator (except fulvestrant for which a washout of at least 6 weeks is required).
* Inadequate hematological function.
* Inadequate renal function with serum creatinine ≥1.5 x upper limit of normal (ULN).
* Liver function: aspartate aminotransferase >3 x ULN, or alanine aminotransferase >3 x ULN. Total bilirubin >1.5 x ULN.
* Non-resolution of any prior treatment related toxicity to <Grade 2, except for alopecia

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-10-27 (Actual); Study Completion 2024-12-26 (Actual)

PRIMARY OUTCOMES:
Investigational medicinal product (IMP)-related dose limiting toxicities (DLTs) | Day 1 to Day 28
  Incidence rate of study treatment-related DLTs at Cycle 1

SECONDARY OUTCOMES:
Safety: Adverse Events (AEs) | Up to 30 days after administration of study treatment
  Number of adverse events related to study therapy
Assessment of Pharmacokinetic parameter of SAR439859: tlag | Day 1 and Day 22 of Cycle 1 (28 days)
  Lag time, interval between administration time and the sampling time preceding the first concentration above the lower limit of quantification
Assessment of Pharmacokinetic parameter of SAR439859: tmax | Day 1 and Day 22 of Cycle 1 (28 days)
  First time to reach Cmax
Assessment of Pharmacokinetic parameter of SAR439859: Cmax | Day 1 and Day 22 of Cycle 1 (28 days)
  Maximum concentration observed
Assessment of Pharmacokinetic parameter of SAR439859: AUC0-24h or AUC0-10h and/or AUC0-12h | Day 1 and Day 22 of Cycle 1 (28 days)
  Area under the plasma concentration versus time curve over the dosing interval (24 hours, 10 hours or 12 hours)
Assessment of Pharmacokinetic parameter of SAR439859: Ctrough | Day 1, Day 8, Day 15 and Day 22 of Cycle 1 (28 days) and Day 1 of Cycle 2
  Plasma concentration observed just before treatment administration during repeated dosing
Assessment of antitumor activity: Objective response rate (ORR) | 64 weeks
  Objective response rate (ORR) as per Response Evaluation Criteria in Solid Tumors (RECIST 1.1)
Assessment of antitumor activity: Clinical benefit rate (CBR) | 64 weeks
  Clinical benefit rate is (CR [complete response] +PR [partial response] +SD [stable disease] ≥24 weeks) as per RECIST 1.1
Assessment of antitumor activity: Duration of response | 64 weeks
  Response duration defined as the time from initial response to the first documented tumor progression
Assessment of antitumor activity: Non-progression rate | 64 weeks
  Non-progression rate at 24 weeks (percentage of participants without progression at 24 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- Japan (3):
  - Investigational Site Number : 3920003, Nagoya, Aichi-ken
  - Investigational Site Number : 3920001, Kashiwa-shi, Chiba
  - Investigational Site Number : 3920002, Chuo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Tamura K, Mukohara T, Yonemori K, Kawabata Y, Nicolas X, Tanaka T, Iwata H. Phase 1 study of oral selective estrogen receptor degrader (SERD) amcenestrant (SAR439859), in Japanese women with ER-positive and HER2-negative advanced breast cancer (AMEERA-2). Breast Cancer. 2023 May;30(3):506-517. doi: 10.1007/s12282-023-01443-8. Epub 2023 Mar 29. PMID 36977973
- See also: TED15954 Plain language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25357&tenant=MT_SNY_9011